CLINICAL TRIAL: NCT03925831
Title: The Trend Analysis and Associated Factors of Initiating the Service of Pediatric Palliative Care
Brief Title: Trend Analysis of the Service of Pediatric Palliative Care
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201902014RINA
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-02

CONDITIONS: Nursing Caries; Palliative Care; Pediatric Population; Pediatric Cancer; Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Palliative care has received considerable attention in Taiwan in recent years. The relevant research has been widely conducted for palliative care in adult population. However, the research in children population is relatively insufficient. In the limited studies, most of them are the experiences generated from individual institutions. This study is going to retrieve the data from 2008-2017 National Health Insurance Research Database, Cancer Registry Database, Death Registry Database and other relevant materials in order to analyze the trends of using pediatric palliative care service, the types of services, the timing of initiating palliative care, and the preference of using palliative care service among different life span in the past decade. In addition, the study will examine the differences of the timing of initiating of pediatric palliative care service and the types of diseases among different characteristics of children and healthcare providers. And the study will discuss how pediatric palliative care services affect medical costs.

ELIGIBILITY:
Inclusion Criteria:

Individuals died from cancer between 2008 and 2017.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals died from cancer in the National Health Insurance Database.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Taiwan Health and Welfare Data | 2008-2017
  The study will use the National Health Insurance Database, Cancer Registry Database and other relevant materials from Ministry of Health and Welfare in Taiwan to conduct research.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Universtiy Hospital, Taipei, Taiwan